CLINICAL TRIAL: NCT04060589
Title: A Prospective Cohort Study in Men With a Suspicion of Prostate Cancer Who Are Referred Onto an MRI-based Diagnostic Pathway With Donation of Tissue, Blood and Urine for Biomarker Analyses (ReIMAGINE Prostate Cancer Risk)
Brief Title: ReIMAGINE Prostate Cancer Risk
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government); Cancer Research UK (Other); Imperial College London (Other); King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 123973
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Magnetic resonance imaging-targeted biopsy; Biomarker; MRI-based diagnostic pathway; magnetic resonance imaging; targeted biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tissue and Organ Procurement; Blood Donation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort Observation: This is a cohort study where participating men will be asked to donate blood, urine, tissue in addition to access to standard of care tissue and medical data (including imaging files). Men will also consent to longer term healthcare data linkage.
  Interventions: Other: Tissue donation; Other: Blood Donation; Other: Urine Donation; Other: Healthcare data linkage

INTERVENTIONS:
Other: Tissue donation — Biopsies will be performed as part of standard of care, additional cores will be performed for research. Access to standard of care prostate biopsy tissue will also be requested after standard of care reporting is complete.
Other: Blood Donation — Phlebotomy will be performed prior to tissue collection following trust standard operating procedures or drawn when cannula already in situ in preparation for the prostate biopsy.
Other: Urine Donation — Urine will be collected prior to prostate biopsy
Other: Healthcare data linkage — Men will consent to healthcare data linkage via national databases.

SUMMARY:
ReIMAGINE Prostate Cancer Risk is a multi-centre, prospective, observational, longitudinal cohort study of men referred to secondary care with a suspicion of prostate cancer. The aim of the study is to develop a robust baseline risk stratification system for men at risk of prostate cancer.

Men whose serum Prostate Specific Antigen (PSA) level is 20ng/ml or less, whose multi-parametric magnetic resonance imaging (mpMRI) scan has been scored as Prostate Imaging Reporting and Data System (PIRADS)/LIKERT score 3, 4 or 5, and who have been advised and accepted the need for a targeted and systematic prostate biopsy will be invited to take part in the study and be asked to donate blood, urine, imaging files and prostate biopsy for biomarker analysis.

DETAILED DESCRIPTION:
ReIMAGINE Prostate Cancer Risk is a multi-centre, prospective, observational, longitudinal cohort study of men referred to secondary care with a suspicion of prostate cancer or men who are undergoing further tests for prostate cancer staging assessment. Men with a serum PSA level of 20ng/ml or less, whose mpMRI scan has been scored as PIRADS/LIKERT score 3, 4 or 5, and who have been advised and accepted the need for a targeted and systematic prostate biopsy will be invited to enrol.

Men will be recruited across a number of high-volume National Health Service (NHS) centres which already have an mpMRI based diagnostic pathway. All eligible patients referred to secondary care with a suspicion on prostate cancer will be considered for screening. Potential participants will be identified at the point of referral or routine urology cancer clinics. Patients will be approached by the ReIMAGINE study team and consented. The initial discussion may be over the telephone Once the consent form is signed, patients will be asked to donate blood, urine and three additional samples of prostate tissue (taken at the time of their biopsy) for biomarker and Deoxyribonucleic acid (DNA) analysis.

Imaging files from the MRI scan will also be collected and stored on the study data warehouse. Small sections of tissue will be cut from the standard of care blocks (post NHS reporting) and then returned back to the hospital.

After collection of the cross-sectional biological samples within ReIMAGINE, men will revert to NHS standard of care, attending a routine outpatient appointment to obtain the results from their biopsy. We will collect healthcare information on study participants during the study and three years after their prostate biopsy. Further funding will be explored for life-long collection of this data.

The ReIMAGINE team aim to recruit 1,000 men with a PIRADs/LIKERT score 3, 4 or 5 who are undergoing an MRI-directed prostate biopsy. Of these 1,000 biopsies, we anticipate that 60% will have any cancer detected on histology (3+3 or greater) giving approximately 400 cases of clinically significant cancer (Gleason 7 or more).

ELIGIBILITY:
Inclusion Criteria:

* Any man with PSA 20 or less (value recorded <90 days before study entry)
* Men who have undergone a prostate MRI as a standard NHS diagnostic work-up
* MRI lesion conforming to Likert/PIRADS 3, 4 or 5
* Radiological stage T3b or less
* Clinical or radiological stage N0 and M0
* No anti-androgen exposure in the preceding 6 months (5-alpha reductase inhibitors permitted)
* No prior treatment for prostate cancer (chemical, biological, ablative, surgical, radiotherapy)
* Previous trans urethral resection of the prostate (TURP) is permitted
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Men unable to donate tissue, blood or urine.
* Previous prostate cancer treatment
* Previous prostate biopsy <12 months from date of the mpMRI scan used to assess study eligibility (scoring PIRADS/Likert 3, 4 or 5)

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who have been referred to secondary care with a suspicion of prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Presence of clinically significant prostate cancer confirmed on biopsy, defined as any Gleason pattern 7 or greater | 6 weeks
  Proportion of men with significant prostate cancer categorised as gleason pattern 7 or greater
Time to metastases in men with prostate cancer | 3 years
  Development of secondary cancers or cancer recurrence
Time to prostate cancer related death | 3 years
  Time to prostate cancer related death in men diagnosed with prostate cancer

SECONDARY OUTCOMES:
Time to new prostate cancer in men without cancer at baseline | 3 years
  Presence of newly diagnosed prostate cancer in men who were cancer free at baseline
Time to cancer progression in men identified with prostate cancer at baseline | 3 years
  Time to cancer progression in men identified with prostate cancer at baseline
Time to prostate cancer specific death in all men | 3 years
  Time to prostate cancer specific death in all men
Time to all-cause death in all men | 3 years
  Time to all-cause death in all men

CONTACTS AND LOCATIONS:
Overall Officials: Hashim U Ahmed, FRCS, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - University College London Hospital, London
  - Royal Free Hospital, London
  - Charing Cross Hospital, London

REFERENCES:
- [Derived] Marsden T, Ahmed HU, Emberton M; ReIMAGINE Study Group. An update from the ReIMAGINE Prostate Cancer Risk Study (NCT04060589): A prospective cohort study in men with a suspicion of prostate cancer who are referred onto a magnetic resonance imaging-based diagnostic pathway with donation of tissue, blood, and urine for biomarker analyses. Eur Urol. 2021 Oct;80(4):398-399. doi: 10.1016/j.eururo.2021.06.011. Epub 2021 Jul 1. PMID 34218972